CLINICAL TRIAL: NCT06920173
Title: The PULSE Study - The Peripheral Use of Low-dose Vasopressors for Safety and Efficacy in the Intensive Care Unit: a Pilot Feasibility Study
Brief Title: Pulse Study: Peripheral Use of Low-dose Vasopressors for Safety and Efficacy in the Intensive Care Unit
Acronym: PULSE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Kingston Health Sciences Centre (Other)
Responsible Party: Principal Investigator, Dr. Gordon Boyd, Associate Professor, Kingston Health Sciences Centre
Organization: Queen's University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 6042888
Record Dates: First submitted 2025-03-04; First posted 2025-04-09 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Shock; Peripheral Venous Catheterization; Central Venous Catheterization; Critically Ill Patients Admitted in ICU
Keywords: critical illness; peripheral vasopressor use; intensive care unit; feasibility study; peripheral venous catheter; central venous catheter
MeSH Terms: conditions — Shock; Critical Illness

STUDY DESIGN:
Intervention Model Description: The proposed study design is a prospective, pragmatic, unblinded feasibility study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Peripheral Venous Catheter (Experimental): Patients in this arm will have vasopressors infusing through a peripheral venous catheter. If patients have escalating doses of vasopressors or require more than 2 vasopressors, they will have a central venous catheter placed.
  Interventions: Procedure: Experiemental: Peripheral Venous Catheter
- Central Venous Catheter (Active Comparator): Patients in this group will have vasopressors infusing through a central venous catheter
  Interventions: Procedure: Experiemental: Peripheral Venous Catheter

INTERVENTIONS:
Procedure: Experiemental: Peripheral Venous Catheter — Patients older than 18 years of age who present with shock requiring vasopressors at the following minimum doses: norepinephrine 5 mcg/min, phenylephrine 50 mcg/min, epinephrine 5 mc/min, dobutamine 5 mcg/kg/min. Vasopressors are infused through a peripheral venous catheter (18 gauge or larger); however, patients are crossed over to the central venous catheter group if the maximum vasopressor dose is reached or more than two vasopressors.

SUMMARY:
Using medications to increase blood pressure, called vasopressors, is invaluable in treating patients who have difficulty maintaining stable blood pressure. Vasopressors are usually infused through a central venous catheter (CVC), which is a flexible tube placed in the large vein of the neck, arm or groin. CVCs require a skilled clinician and often with an ultrasound to prevent complications such as a collapsed lung or bleeding. Alternatively, the infusion of vasopressors through a peripheral venous catheter (PVC), a thin tube placed in the smaller veins of the arm or hand has been avoided due to the risk of extravasation, which is the leakage of fluid to surrounding tissues. This can lead to potential tissue death requiring surgery. However, emerging research shows the safety of infusing vasopressors through a PVC, referred to as peripheral vasopressors. There is a growing interest in peripheral vasopressors for two main reasons: to expedite vasopressor initiation in patients with refractory shock and to avoid CVC placement and its potential complications. However, a standardized protocol for administration is lacking and many clinicians still avoid peripheral vasopressors due to lack of high-quality evidence. The investigators will examine the effectiveness of implementing a peripheral vasopressor protocol by conducting a feasibility study and assessing outcomes such as the safety of peripheral vasopressors and the acceptability rate of healthcare providers. By conducting this study, the investigators aim to provide the framework to conduct larger, multi-center trials and to provide high-quality data for the future use of a standardized peripheral vasopressor protocol.

DETAILED DESCRIPTION:
In the intensive care unit (ICU), vasopressors are administered when fluid resuscitation alone cannot maintain adequate blood pressure in patients with shock. The standard of care for continuous infusions of vasopressors is through a central venous catheter (CVC) rather than a peripheral venous catheter (PVC). The use of CVCs prevents extravasation, which can lead to local tissue ischemia resulting in necrosis. However, CVC placement is not a benign procedure requiring a skilled clinician and the use of ultrasound guidance to prevent complications such as pneumothorax, bleeding or erroneous arterial cannulation. Furthermore, complications related to the maintenance of CVCs include deep vein thrombosis (DVT), and central line-associated blood stream infections (CLABSIs). These recognized complications occur in more than 15% of patients. There is a growing interest in peripheral vasopressor use for two main reasons: to expedite vasopressor administration in patients with refractory shock and to potentially avoid CVC placement and it complications. However, there remains no standardized protocols and many clinicians still believe that vasopressors must be infused through a CVC despite current evidence showing the safety of peripheral vasopressors. However, to date only observational studies have been performed. A randomized control trial is needed to provide high quality data to improve the future use of peripheral vasopressors, which has the potential to positively impact patient care.

The investigators will perform a feasibility study for the implementation of a peripheral vasopressor protocol. They will also assess the safety of the peripheral vasopressor protocol and evaluate clinically relevant outcomes, which will be listed below. The investigators hypothesize that implementing a peripheral vasopressor protocol is feasible and safe.

Aim 1: Adapt a peripheral vasopressor protocol and perform a feasibility study. The investigators will conduct a feasibility study to determine the efficacy of a peripheral vasopressor protocol. In collaboration with an ICU pharmacist, the investigators will adopt a peripheral vasopressor protocol at Kingston Health Sciences Center to determine the dosages and concentrations of each vasopressor. The participants will be randomized 1:1:1 into a low-dose peripheral vasopressor group vs. a dose peripheral vasopressor group vs a high-dose peripheral vasopressor group vs a CVC group. Based on the admission rates of our ICU, the investigators aim to recruit 25 patients into each group. They will investigate the feasibility of recruitment, data capture rate, acceptability rate by nursing staff and providers of the peripheral vasopressor protocol and avoidance rate of CVC placement.

Aim 2a: Perform a safety assessment of peripheral vasopressor protocol. The investigators will assess the safety of peripheral vasopressor administration after two months of protocol initiation. Specific adverse events to be captured include extravasation (+/- tissue necrosis), pneumothorax, arterial cannulation, and deep vein thrombosis. The investigators will assess any differences in adverse events between the low-dose peripheral vasopressor group vs the high-dose peripheral vasopressor group vs the CVC group, which will be reported as proportions. The investigators hypothesize that peripheral vasopressor use will be safe compared to the CVC group, with few to no adverse events.

Aim 2b: Determine the impact of a peripheral vasopressor protocol on clinically relevant outcomes. This feasibility study will investigate secondary outcomes such as alive and central line-free days, infection rates including CLABSIs, mortality and ICU/hospital length of stay. The investigators will report these outcomes as medians with 95% confidence intervals.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 or older who do not have a central line or PICC line already placed
* Presence of shock requiring vasopressors at the following minimum doses: norepinephrine 5 mcg/min, phenylephrine 50 mcg/min, epinephrine 5 mc/min, dobutamine 5 mcg/kg/min

Exclusion Criteria:

* Urgent need for dialysis requiring placement of hemodialysis catheter
* More than two vasopressors are required to maintain a MAP >65 on admission to the ICU
* Pregnancy or suspected pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-02-03 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
The feasibility of recruitment | 1 week
  We hope to recruit at least 80% of patients who are eligible for the study.
Feasibility of data capture rate | 1 week
  We hope to have a data capture rate of at least 90%
Feasibility of acceptability rate of peripheral vasopressor protocol | 1 week
  We hope to have an acceptability rate of at least 90% by providers and nurses

SECONDARY OUTCOMES:
Avoidance of central venous catheter placement | 1 week
  We will evaluate the crossover rate in patients who are initiated on peripheral vasopressors but ultimately require a central line due to escalating doses of vasopressors or poor venous access. We hope that 50% of patients will need a central line who have been initially allocated to the PVC group.
Assessing extravasation rates | 1 week
  This will be reported using descriptive statistics with a confidence interval of 95%.
Assessing alive and central line-free days | 1 week
  This will be reported as medians with a 95% confidence interval.
Assessing central-line associated blood stream infections | 1 week
  This will be reported as medians with a 95% confidence interval.
Assessing mortality rate | 1 week
  This will be reported as medians with a 95% confidence interval.
Assessing ICU and hospital length of stay | 1 week
  This will be reported as medians with a 95% confidence interval.

CONTACTS AND LOCATIONS:
Overall Officials: Gord Dr., PhD, MD, Principal Investigator — Queen's University, Kingston Health Sciences Center
Locations (1):
- Kingston Health Sciences Center, Kingston, Ontario, Canada

IPD SHARING:
Plan to Share IPD: Yes
Data that will be shared include age, sex, admission date and admitting diagnosis, peripheral IV location and gauge, vasopressor type, duration of vasopressor and complications.

REFERENCES:
- [Background] Marti K, Hartley C, Sweeney E, Mah J, Pugliese N. Evaluation of the safety of a novel peripheral vasopressor pilot program and the impact on central line placement in medical and surgical intensive care units. Am J Health Syst Pharm. 2022 Aug 19;79(Suppl 3):S79-S85. doi: 10.1093/ajhp/zxac144. PMID 35605137
- [Background] Loubani OM, Green RS. A systematic review of extravasation and local tissue injury from administration of vasopressors through peripheral intravenous catheters and central venous catheters. J Crit Care. 2015 Jun;30(3):653.e9-17. doi: 10.1016/j.jcrc.2015.01.014. Epub 2015 Jan 22. PMID 25669592
- [Background] Munroe ES, Heath ME, Eteer M, Gershengorn HB, Horowitz JK, Jones J, Kaatz S, Tamae Kakazu M, McLaughlin E, Flanders SA, Prescott HC. Use and Outcomes of Peripheral Vasopressors in Early Sepsis-Induced Hypotension Across Michigan Hospitals: A Retrospective Cohort Study. Chest. 2024 Apr;165(4):847-857. doi: 10.1016/j.chest.2023.10.027. Epub 2023 Oct 26. PMID 37898185
- [Background] McGee DC, Gould MK. Preventing complications of central venous catheterization. N Engl J Med. 2003 Mar 20;348(12):1123-33. doi: 10.1056/NEJMra011883. No abstract available. PMID 12646670
- [Background] Stolz A, Efendy R, Apte Y, Craswell A, Lin F, Ramanan M. Safety and efficacy of peripheral versus centrally administered vasopressor infusion: A single-centre retrospective observational study. Aust Crit Care. 2022 Sep;35(5):506-511. doi: 10.1016/j.aucc.2021.08.005. Epub 2021 Sep 30. PMID 34600834
- [Background] Kalinoski M, Kalinoski T, Pendleton K. The use of peripheral vasopressors and its implications for hospital medicine. Br J Hosp Med (Lond). 2024 Jul 30;85(7):1-8. doi: 10.12968/hmed.2024.0048. Epub 2024 Jul 24. PMID 39078910
- [Background] Abu Sardaneh A, Penm J, Oliver M, Gattas D, McLachlan AJ, James C, Cella C, Aljuhani O, Acquisto NM, Patanwala AE. International pharmacy survey of peripheral vasopressor infusions in critical care (INFUSE). J Crit Care. 2023 Dec;78:154376. doi: 10.1016/j.jcrc.2023.154376. Epub 2023 Aug 2. PMID 37536012
- [Background] Owen VS, Rosgen BK, Cherak SJ, Ferland A, Stelfox HT, Fiest KM, Niven DJ. Adverse events associated with administration of vasopressor medications through a peripheral intravenous catheter: a systematic review and meta-analysis. Crit Care. 2021 Apr 16;25(1):146. doi: 10.1186/s13054-021-03553-1. PMID 33863361
- [Background] Yerke JR, Mireles-Cabodevila E, Chen AY, Bass SN, Reddy AJ, Bauer SR, Kokoczka L, Dugar S, Moghekar A. Peripheral Administration of Norepinephrine: A Prospective Observational Study. Chest. 2024 Feb;165(2):348-355. doi: 10.1016/j.chest.2023.08.019. Epub 2023 Aug 21. PMID 37611862